CLINICAL TRIAL: NCT00758069
Title: Phase II Study on Sitagliptin -Assessment of Glucose-lowering Effects
Brief Title: Clinical Study on Sitagliptin for Assessment of Glucose-lowering Effects (0431-045)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-045; MK0431-045; 2008_026
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo
- 2 (Experimental): Sitagliptin 100 mg
  Interventions: Drug: sitagliptin phosphate
- 3 (Experimental): Sitagliptin 50 mg
  Interventions: Drug: Comparator: Sitagliptin

INTERVENTIONS:
Drug: sitagliptin phosphate — 100 mg once daily (QD), taken orally for 4 weeks
  Other Names: MK0431
  Arms: 2
Drug: Comparator: Placebo — Placebo tablet, QD, taken orally for 4 weeks
  Arms: 1
Drug: Comparator: Sitagliptin — 50 mg twice daily (BID), taken orally for 4 weeks
  Other Names: MK0431
  Arms: 3

SUMMARY:
A clinical study determines the safety and efficacy of sitagliptin (MK0431) in patients with Type 2 diabetes mellitus who have inadequate glycemic control on diet/exercise therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients Have Type 2 Diabetes Mellitus On Diet/Exercise Therapy

Exclusion Criteria:

* Patients Have Type 1 Diabetes Mellitus

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-07-03 (Actual); Primary Completion 2006-02-13 (Actual); Study Completion 2006-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Nonaka K, Tsubouchi H, Okuyama K, Fukao Y, Johnson-Levonas AO, Amatruda JM. Effects of once-daily sitagliptin on 24-h glucose control following 4 weeks of treatment in Japanese patients with type 2 diabetes mellitus. Horm Metab Res. 2009 Mar;41(3):232-7. doi: 10.1055/s-0028-1100413. Epub 2009 Feb 27. PMID 19253204
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase II.
  First patient in: 31 July 2005. Last patient, last visit: 13 February 2006.
  The study was conducted at 8 centers in Japan.
Pre-assignment Details: Patients 20-69 years of age with type 2 diabetes mellitus and inadequate glycemic control (HbA1c ≥6.5% and <10% at Week -2) were eligible for randomization following at least 8 weeks of diet/exercise and antihyperglycemic agent (AHA) wash-off (for patients previously on an AHA), including a 2-week placebo run-in.
Groups:
- Sitagliptin 100 mg QD: The Sitagliptin 100 mg QD group includes data from all patients randomized to receive treatment with sitagliptin 100 mg orally once daily (QD=once daily).
- Sitagliptin 50 mg BID: The Sitagliptin 50 mg BID group includes data from all patients randomized to receive treatment with sitagliptin 50 mg orally twice daily (BID=twice daily).
- Placebo: The Placebo group includes data from all patients randomized to receive treatment with matching placebo orally.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo
Started | 27 (Study enrolled slightly more than the target of N=20) | 25 (Study enrolled slightly more than the target of N=20) | 28 (Study enrolled slightly more than the target of N=20)
Completed | 26 | 25 | 27
Not Completed | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Incorrect Study Drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo | Total
Number analyzed (Participants) | 27 | 25 | 28 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (8.9) | 56.1 (8.9) | 53.6 (10.3) | 54.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 8 | 25
  Male | 17 | 18 | 20 | 55
24-hour weighted mean plasma glucose (24hr-WMG) [Mean (Standard Deviation); unit: mg/dL] — The 24hr-WMG is the weighted mean of the blood glucose weighted by the intervals between time points for a day [i.e. the area under curve in glucose-time profile through 24-hours (AUC0-24 hr) divided by 24].
  mg/dL | 195.0 (55.6) | 188.9 (46.6) | 195.4 (46.2) | 193.2 (49.1)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 158.6 (41.0) | 156.4 (41.3) | 164.1 (36.9) | 159.9 (39.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Weighted Mean Plasma Glucose
Description: Change from baseline at Week 4 is defined as 24-hour weighted mean glucose (24hr-WMG) at Week 4 minus 24hr-WMG at Week 0.
Time Frame: Baseline and Week 4
Population: The Per Protocol population included patients with baseline and Week 4 (i.e., final primary timepoint) values for this outcome and excluded patients who met predefined criteria for protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo
Number analyzed (Participants) | 25 | 24 | 27
mg/dL | -34.9 [-40.9 to 28.9] | -28.6 [-34.7 to 22.4] | -9.0 [-14.8 to -3.2]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustment among the pairwise comparisons of sitagliptin against placebo; ANCOVA model with terms of treatment as a factor and baseline value as a covariate was used for pairwise comparison; Least-squares Mean Difference = -25.9, 95% CI [-34.2 to -17.5] — ANCOVA model with terms of treatment as a factor and baseline value as a covariate was used to estimate difference of two groups and its 95% confidence interval
Statistical Analysis 2: Comparison: Sitagliptin 50 mg BID vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustment among the pairwise comparisons of sitagliptin against placebo; ANCOVA model with terms of treatment as a factor and baseline value as a covariate was used for pairwise comparison; Least-squares Mean Difference = -19.5, 95% CI [-28.0 to -11.1] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Plasma Glucose
Description: Change from baseline at Week 4 is defined as fasting plasma glucose at Week 4 minus fasting plasma glucose at Week 0.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo
Number analyzed (Participants) | 25 | 24 | 27
mg/dL | -22.3 [-27.7 to 17.0] | -16.0 [-21.4 to 10.6] | -3.1 [-8.2 to 2.0]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustment among the pairwise comparisons of sitagliptin against placebo; ANCOVA model with terms of treatment as a factor and baseline value as a covariate was used for pairwise comparison; Least-squares Mean Difference = -19.3, 95% CI [-26.6 to -11.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg BID vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustment among the pairwise comparisons of sitagliptin against placebo; ANCOVA model with terms of treatment as a factor and baseline value as a covariate was used for pairwise comparison; Least-squares Mean Difference = -12.9, 95% CI [-20.4 to -5.4] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 2 | 0
Other Adverse Events (participants affected / at risk) | 1 | 1 | 2
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo
Overdose (Injury, poisoning and procedural complications) | 1/27 | 2/25 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg QD | Sitagliptin 50 mg BID | Placebo
Nasopharyngitis (Infections and infestations) | 1/27 | 1/25 | 2/28

LIMITATIONS AND CAVEATS:
Reported overdoses, regardless of association with reported adverse events, were considered as serious adverse events in this study. The patients for whom the event of overdose was reported had no concomitant AEs with the overdose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.